CLINICAL TRIAL: NCT00584233
Title: Evaluation of Breast CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 214750; 1R01CA181081 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed; Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast CT and Breast MRI (Experimental): Four hundred women who will be having breast biopsy as part of their standard care (BIRADS 4 and 5) will undergo pre- and post- contrast breast computed tomography and pre- and post- contrast magnetic resonance imaging.
  Interventions: Device: computed tomography; Device: MRI

INTERVENTIONS:
Device: computed tomography — Computed tomography of both breasts. For all subjects, CT scanning will be performed before and after an I.V. iodinated contrast injection (100 mL).
  Other Names: Breast x-ray
Device: MRI — Breast MRI

SUMMARY:
The investigators have studied the potential of breast computed tomography (bCT) for breast imaging under an NIH-funded Biomedical Research Partnership (BRP) grant (R01 EB002138-10), and 4 breast CT scanners have been developed that have imaged over 600 women to date (under more than one IRB-approved protocol). The BRP grant cannot be renewed, and with this (resubmitted) R01 grant application, the investigators seek to finalize the investigators' research in breast CT - The specific aims have been significantly modified as a result of the first critique, and the investigators now focus on a narrower set of remaining issues.

This version of the protocol will add breast magnetic resonance imaging (MRI) to the experimental procedures.

DETAILED DESCRIPTION:
Clinical evaluation: Four hundred women who will be having breast biopsy as part of their standard care (BIRADS 4 and 5) will be recruited to undergo additional imaging prior to biopsy, including (research) pre-and post-contrast enhanced breast CT imaging of both breasts, as well as (standard, FDA approved) contrast enhanced breast MRI. The potential of non-contrast enhanced breast CT will be compared using receiver operating characteristic (ROC) methodology against mammography alone, as well as with mammography + tomosynthesis. The breast CT images (including both pre-and post-contrast images) will be compared using ROC methodology against standard-of-care contrast-enhanced MRI (which includes both non-contrast and contrast images). The results of the clinical trials proposed in this investigation should provide strong evidence in regards to the potential of breast CT for breast cancer screening in the normal risk and high risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 35 years old
* Diagnostic findings from prior mammography highly suggestive of breast malignancy (BI- RADS® category 4 or BI-RADS® category 5)
* Not pregnant or breast-feeding
* Ability to lie motionless for up to 5 minutes

Exclusion Criteria:

* Recent breast biopsy
* History of moderate or severe reaction to contrast agent injection
* History of Allergy to Iodine
* History of multiple food and/or drug allergy
* Currently taking Glucophage or Glucovance (Metformin)
* History of Chronic Asthma
* History of Diabetes Mellitus
* Renal (kidney) disease, or solitary kidney
* Recent lab tests showing elevated serum creatinine (≥ 1.5 mg/dL)
* Recent lab tests showing estimated glomerular filtration rate (eGFR) ≤ 60 ml/minute
* Positive urine pregnancy test or currently breast-feeding
* Inability to understand the risks and benefits of the study
* The standard MRI contraindications apply, including but not limited to: having a pacemaker or other implanted electronic device, metal foreign bodies within the eye, aneurysm clips, heart valve prosthesis, vascular stents, coils, intrauterine devices (IUDs), inferior vena cava (IVC) filters, gunshot wounds with retained bullet fragments.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-11-22 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Boone, Ph.D., Principal Investigator — UC Davis Dept. of Radiology
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breast CT and Breast MRI
Started | 75
Completed | 57
Not Completed | 18
Not completed — Withdrawal by Subject | 5
Not completed — Subjects did not complete both CT and MRI to be evaluated in results | 13

BASELINE CHARACTERISTICS:
Arm/Group | Breast CT and Breast MRI
Number analyzed (Participants) | 57
Age, Continuous [Geometric Mean (Full Range); unit: years] | 57 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 45
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Pre- and Post- Contrast Breast Computed Tomography With Pre- and Post- Contrast Magnetic Resonance Imaging.
Description: The specific quantitative endpoint of the analysis is the difference in area under the receiver operating characteristic curve (AUC) between contrast-enhanced breast CT (CE-bCT) and contrast-enhanced breast MRI (CE-bMRI).
Time Frame: 5 years
Population: The analysis patient population includes women characterized as BIRAD's 4 and 5 patients based upon screening mammography (or tomosynthesis), who will then undergo further imaging workup based upon a positive finding on screening mammography (or tomosynthesis) or a palpable lesion. Because these women will be having a breast needle core biopsy after imaging, the lesion histopathology will be known and we can classify patients as having either benign or malignant lesions.
Measure: Mean (Standard Error); unit: probability
Arm/Group | Breast CT and Breast MRI
Number analyzed (Participants) | 57
probability | -0.04 (0.02)
Statistical Analysis 1: Comparison: Breast CT and Breast MRI; The analysis is intended to evaluate non-inferiority in observer performance between CE-bCT and CE-bMRI as assessed by the area under the ROC curve (AUC). The null hypothesis is that the observed difference in average AUC for CE-bCT and CE-bMRI will be outside of a non-inferiority margin of -0.04. See below for details of the power analyses; Test type: Non-Inferiority — The statistical test will be to assess non-inferiority. The non-inferiority margin is -0.04 in AUC. Key parameters are the number of participating patients, the number of radiologists reading the images in the study. Power analysis was conducted using the standard simulation from the ROC literature (Roe and Metz, Academic Radiology 1997). With a total of 100 participating patients and 4 participating readers, we achieve a power >80% with a non-inferiority margin of -0.04; p = 0.05, Obuchowski Rockette; Obuchowski Rockette methodology = 0.05, 95% CI 2-sided [.025 to .975]

ADVERSE EVENTS:
Time Frame: AEs were collected through the course of study activities (up to 21 days). After last study activity was completed, the subject was off study.
Description: Definition does not differ
Arm/Group | Breast CT and Breast MRI
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT00584233/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT00584233/ICF_002.pdf